CLINICAL TRIAL: NCT05898867
Title: Cognitive Bias and Heuristics in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Other Study IDs: CHIPS
Record Dates: First submitted 2023-05-10; First posted 2023-06-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders: Participants from the trial "Reinforcement of Treatment Response in Knee Osteoarthritis: A Randomised Trial" will be defined as responders if they belong to the upper quartile of the change to the pain Visual Analogue Scale (VAS) (those who had the greatest positive changes)
  Interventions: Other: Saline
- Non-responders: Participants from the trial "Reinforcement of Treatment Response in Knee Osteoarthritis: A Randomised Trial" will be defined as non-responders if they belong to the lower quartile of the change to the pain Visual Analogue Scale (VAS) (those who had the smallest change).
  Interventions: Other: Saline

INTERVENTIONS:
Other: Saline — Open label intra-articular injection of isotonic saline.

SUMMARY:
This study aims to understand if certain cognitive biases and heuristics are present in patients with knee osteoarthritis being treated with open label placebo (saline injections in the knee). A predefined survey will investigate the affect heuristic and group interviews patients who have responded well or not so well respectively will be used to examine if other cognitive biases or heuristics are present.

Cognitive biases are systematic patterns of deviation from norm or rationality in judgment, while heuristics are tactics, or mental shortcuts to aid in the decision-making process.

DETAILED DESCRIPTION:
Cognitive biases (systematic patterns of deviation from norm or rationality in judgment) and heuristics (tactics, or mental shortcuts to aid in the decision-making process) are increasingly being used in healthcare to facilitate good health decisions, improved care, and in designing new interventions.It has also been shown that cognitive biases influence how patients rate their own health.

Less is known about which specific cognitive biases and/or heuristics that are in play when patients with knee osteoarthritis form their treatment expectations and evaluate their health following an intervention.

This study aims to understand if certain cognitive biases and heuristics are present in patients with knee (OA) being treated with open label intra-articular placebo injections.

Understanding which cognitive biases and/or heuristics that are in play when these patients evaluate their health outcome following open label placebo, allows future treatment context to be designed in a way that actively utilises these cognitive biases and/or heuristics to obtain a greater magnitude of response.

A global predefined questionnaire, evaluating the presence and strength of the affect heuristic, is sent to all participants from the study "Reinforcement of Treatment Response in Knee Osteoarthritis: A Randomised Trial" (Clinical trial.gov registration: NCT05225480). In addition investigators will invite responders and non-responders respectively from the same study to group interviews in order to produce a structured conceptualisation map; the group content mapping method.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in the study "Reinforcement of Treatment Response in Knee Osteoarthritis: A Randomised Trial" (Clinical trial.gov registration: NCT05225480)

Exclusion Criteria:

* Have not participated in the study "Reinforcement of Treatment Response in Knee Osteoarthritis: A Randomised Trial" (Clinical trial.gov registration: NCT05225480)

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People over 50 years of age with tibiofemoral knee osteoarthritis according to the American College of Rheumatology with an average knee pain in the last week during weight bearing activities of at least 4 on a 0 to 10 points VAS scale (0=no pain; 10=worst possible pain).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Concept maps. | The GCM sessions are carried out approximately 1 year and 2 months after baseline.
  Using the Group Concept Mapping (GCM) method investigators will generate concept maps from non-responders and responders respectively, from participants from the study "Reinforcement of Treatment Response in Knee Osteoarthritis: A Randomised Trial" (Clinical trial.gov registration: NCT05225480)
  Responders are defined as the those patients that had the largest change (4th quartile) to the pain Visual Analog Scale (VAS) (0-100mm). Non-responders are defined as the 1st quartile (least change).
  GCM is a formal group process using a structured approach to identify ideas on a topic of interest and organise them into domains based on a mixed-method participatory design that incorporates group processes and multivariate statistical analyses (multidimensional scaling and hierarchical cluster analysis).
  Using the concept maps and statements, investigators will assess similarities with known cognitive biases or heuristics.

SECONDARY OUTCOMES:
Strength of the affect heuristic in patients with knee OA | The questionnaire is administered approximately 1 year and 4 months after baseline.
  Using a questionnaire tool investigators will asses the strength of the affect heuristic with participants from from the study "Reinforcement of Treatment Response in Knee Osteoarthritis: A Randomised Trial" (Clinical trial.gov registration: NCT05225480).
  The strength of the affect heuristic is expressed via the correlation coefficient which ranges from (-1 to 1) and the 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg-Frederiksberg Hospital, Copenhagen, Denmark

DOCUMENTS (1):
  • Study Protocol (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT05898867/Prot_000.pdf